CLINICAL TRIAL: NCT01527357
Title: A Phase 3, Randomized, Single-blind, Controlled Trial of Topical Fibrocaps™ in Intraoperative Surgical Hemostasis
Brief Title: A Study of Fibrocaps™ in Surgical Bleeding
Acronym: FINISH-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FC-004
Record Dates: First submitted 2012-01-26; First posted 2012-02-07 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2016-07

CONDITIONS: Mild or Moderate Surgical Bleeding
Keywords: fibrin sealant; thrombin; fibrinogen; hemostasis
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Fibrin Tissue Adhesive; Gelatin Sponge, Absorbable; Fibrin Foam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibrocaps + Gelatin Sponge (Experimental): Single application of Fibrocaps plus gelatin sponge.
  Interventions: Biological: Fibrocaps; Biological: Gelatin sponge
- Gelatin Sponge (Active Comparator): Single application of gelatin sponge alone.
  Interventions: Biological: Gelatin sponge

INTERVENTIONS:
Biological: Fibrocaps — Human fibrinogen and thrombin powder, for topical administration.
  Other Names: PRO-0601; Fibrin sealant
  Arms: Fibrocaps + Gelatin Sponge
Biological: Gelatin sponge — Absorbable gelatin sponge for topical administration.
  Other Names: Gelfoam; Spongostan

SUMMARY:
The purpose of this study is to confirm the superiority of Fibrocaps plus gelatin sponge, as compared to gelatin sponge alone, for achieving hemostasis.

The investigational products were used in participants with mild to moderate surgical bleeding during spine, liver, vascular or soft tissue surgery, when control of mild to moderate bleeding by standard surgical techniques is ineffective and/or impractical.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed an institutional review board/independent ethics committee (IRB/IEC)-approved informed consent document
2. Is undergoing one of the 4 surgical procedures described
3. Is at least 18 years old at time of consent
4. If female and of child-bearing potential, has negative pregnancy test during screening and is not breast-feeding
5. If able to reproduce, agrees to use a medically accepted form of contraception from the time of consent to completion of all follow-up study visits when engaging in heterosexual intercourse
6. Has not received blood transfusion between screening and study treatment
7. Has mild to moderate surgical bleeding
8. Does not have intra-operative complications
9. Has not used a topical hemostat containing thrombin prior to study treatment
10. Has an approximate bleeding site surface area of less than or equal to 100 cm^2

Exclusion Criteria:

1. Has known antibodies or hypersensitivity to thrombin or other coagulation factors
2. Has history of heparin-induced thrombocytopenia (only for vascular subjects where heparin use is required)
3. Has known allergy to gelatin sponge
4. Is unwilling to receive blood products
5. Has liver enzymes appropriate for the study, considering their disease
6. Has appropriate level of platelets per liter (PLT/L) during screening
7. Has any clinically-significant coagulation disorder that may interfere with the assessment of efficacy or pose a safety risk to the subject according to the Investigator, or baseline abnormalities during screening that are not explained by current drug treatment (e.g., warfarin, heparin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 721 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2013-04-24 (Actual); Study Completion 2013-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (48):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cardio-Thoracic Surgeons, PC, Birmingham, Alabama
  - University of Southern California, Keck School of Medicine, Los Angeles, California
  - University of Southern California/Norris Comprehensive Cancer Center, Los Angeles, California
  - Vascular Interventional Specialists of Orange County, Orange, California
  - Lotus Clinical Research, LLC, Pasadena, California
  - Boulder Neurological Institute, Boulder, Colorado
  - Spine Colorado, Durango, Colorado
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Bluegrass Orthopedics, Lexington, Kentucky
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Borgess Research Institute, Kalamazoo, Michigan
  - Beaumont Health System, Royal Oak, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - William Muir MD Spine Surgery, Las Vegas, Nevada
  - New York-Presbyterian Hospital/Columbia University, New York, New York
  - Duke University Hospital Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The University of Oklahoma - Tulsa, Tulsa, Oklahoma
  - Oregon Health & Science University Hospital & Clinics, Portland, Oregon
  - University of North Texas Health Sciences Center, Fort Worth, Texas
  - Physician's Research Options, Sandy City, Utah
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Northwest Orthopaedic Specialists, P.S., Spokane, Washington
  - Multicare Neuroscience Center of Washington, Tacoma, Washington
- Belgium (5):
  - Militair Hospitaal Koningin Astrid, Brussells
  - Clinique du Parc Leopold, Service de Neurochirurgie, Brussels
  - Hopital Erasme, Service de Neurochirurgie, Brussels
  - Universitair Ziekenhuis Gent, Gasto-Intestinale Heelkunde, Ghent
  - Universitair Ziekenhuis Leuven, Abdominale Heelkunde, Leuven
- Netherlands (7):
  - Amphia Hospital, Breda
  - Medisch Spectrum Twente, Enschede
  - University Medical Centre Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Rijnstate Arnhem, Velp
- United Kingdom (7):
  - Queen Elizabeth Hospital Birmingham, Birmingham, England
  - Addenbrookes Hospital Vascular Department, Cambridge, England
  - Doncaster Royal Infirmary, Doncaster, England
  - Hull Royal Infirmary, Hull, England
  - Leeds General Infirmary, Leeds, England
  - King's College Hospital, London, England
  - Freeman Hospital, Newcastle upon Tyne, England

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gupta N, Chetter I, Hayes P, O-Yurvati AH, Moneta GL, Shenoy S, Pribble JP, Zuckerman LA. Randomized trial of a dry-powder, fibrin sealant in vascular procedures. J Vasc Surg. 2015 Nov;62(5):1288-95. doi: 10.1016/j.jvs.2015.05.038. Epub 2015 Aug 5. PMID 26254451
- [Derived] Bochicchio GV, Gupta N, Porte RJ, Renkens KL, Pattyn P, Topal B, Troisi RI, Muir W, Chetter I, Gillen DL, Zuckerman LA, Frohna PA. The FINISH-3 trial: a phase 3, international, randomized, single-blind, controlled trial of topical fibrocaps in intraoperative surgical hemostasis. J Am Coll Surg. 2015 Jan;220(1):70-81. doi: 10.1016/j.jamcollsurg.2014.09.019. Epub 2014 Oct 13. PMID 25458801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from May 2012 to April 2013 at 57 investigative sites (United States, n = 28; United Kingdom, n = 12; The Netherlands, n = 11; and Belgium, n = 6), and were randomized 2:1 to receive treatment with Fibrocaps plus gelatin sponge or gelatin sponge alone.
Pre-assignment Details: After screening, 719 eligible participants had surgery in 1 of 4 surgical indications (i.e., spinal, hepatic, vascular, or soft tissue dissection) on Day 1 according to local standard practice, and received treatment with the investigational product assigned.
Period: Overall Study
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Started | 482 | 239
Efficacy Population | 480 (Two participants did not receive study treatment.) | 239
Completed | 465 | 230
Not Completed | 17 | 9
Not completed — Death | 8 | 2
Not completed — Lost to Follow-up | 6 | 4
Not completed — Withdrew Consent | 1 | 1
Not completed — Non-compliance | 0 | 1
Not completed — No Day 29 Visit | 0 | 1
Not completed — Did Not Receive Treatment | 2 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge | Total
Number analyzed (Participants) | 482 | 239 | 721
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (14.44) | 58.1 (14.12) | 57.6 (14.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 115 | 329
  Male | 268 | 124 | 392
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 8 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 20 | 62
  White | 422 | 210 | 632
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis (TTH) for Participants Receiving Spinal Surgery
Description: The measurement of TTH begins at t=0, which is the time the study product is applied to the Target Bleeding Site (TBS) and ends when hemostasis is achieved or 5-minutes, whichever occurs first, based on data collected by surgery type and treatment.
Time Frame: Within 5 minutes
Population: Efficacy population consists of all participants who were randomized, received study treatment, and had a TTH assessment. Number analyzed is the number of participants in the efficacy population who receive each type of surgery.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 122 | 61
minutes | 1.0 [0.5 to 1.5] | 2.5 [1.5 to 4.0]
Statistical Analysis 1: Comparison: Fibrocaps + Gelatin Sponge vs Gelatin Sponge; Test type: Superiority; p < 0.0001, Log Rank

2. Primary Outcome: Time to Hemostasis (TTH) for Participants Receiving Vascular Surgery
Description: as for outcome 1
Time Frame: Within 5 minutes
Population: Efficacy population
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 117 | 58
minutes | 2.0 [1.50 to 2.50] | 4.0 [3.00 to 5.00]
Statistical Analysis 1: Comparison: Fibrocaps + Gelatin Sponge vs Gelatin Sponge; Test type: Superiority; p < 0.0001, Log Rank

3. Primary Outcome: Time to Hemostasis (TTH) for Participants Receiving Hepatic Resection
Description: as for outcome 1
Time Frame: Within 5 minutes
Population: Efficacy population
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 119 | 61
minutes | 1.0 [1.00 to 1.50] | 2.0 [1.50 to 2.50]
Statistical Analysis 1: Comparison: Fibrocaps + Gelatin Sponge vs Gelatin Sponge; Test type: Superiority; p < 0.0001, Log Rank

4. Primary Outcome: Time to Hemostasis (TTH) for Participants Receiving Soft Tissue Dissection
Description: as for outcome 1
Time Frame: Within 5 minutes
Population: Efficacy population
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 122 | 59
minutes | 1.5 [1.00 to 1.50] | 2.5 [2.00 to 3.50]
Statistical Analysis 1: Comparison: Fibrocaps + Gelatin Sponge vs Gelatin Sponge; Test type: Superiority; p < 0.0001, Log Rank

5. Secondary Outcome: Restricted Mean TTH
Description: Restricted mean TTH over 5 minutes is computed using Irwin's estimator, based on data collected by surgery type and treatment.
Time Frame: Within 5 minutes
Population: Efficacy population. Number analyzed is the number of participants with data available for analysis in each surgery type.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 480 | 239
minutes
  Spinal Surgery: number analyzed (Participants) | 122 | 61
  Spinal Surgery | 1.2 (0.08) | 2.7 (0.19)
  Vascular Surgery: number analyzed (Participants) | 117 | 58
  Vascular Surgery | 2.4 (0.14) | 3.5 (0.2)
  Hepatic Resection: number analyzed (Participants) | 119 | 61
  Hepatic Resection | 1.5 (0.09) | 2.5 (0.21)
  Soft Tissue Dissection: number analyzed (Participants) | 122 | 59
  Soft Tissue Dissection | 1.5 (0.09) | 3.1 (0.19)

6. Secondary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence (including clinically significant changes in laboratory values or other clinical tests) experienced by a participant administered a pharmaceutical product regardless of causal relationship with the treatment. A TEAE is any adverse event reported on the case report form that occurs after start of treatment or any adverse event with a missing start date.
Time Frame: Within 29 days
Population: Safety population, defined as all participants who were randomized and received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 480 | 239
Participants | 426 | 214

7. Secondary Outcome: Number of Participants Who Require Alternative Hemostatic Agents at 5 Minutes
Description: If hemostasis is not achieved within 5 minutes, the treatment is considered to have failed, and the surgeon is to implement additional hemostatic measures.
Time Frame: At 5 minutes
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 480 | 239
Participants | 6 | 7

8. Secondary Outcome: Number of Participants Who Required Red Blood Cells
Description: Red blood cells are defined as including World Health Organization (WHO) DRUG terms of "Blood cells, packed human", "Blood, whole", "Red blood cells", "Red blood cells, concentrated" and "Red blood cells, leucocyte depleted".
Time Frame: Within 29 days
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
Number analyzed (Participants) | 480 | 239
Participants | 40 | 22

ADVERSE EVENTS:
Time Frame: From time of surgery (Day 1) through Day 29 (End of Study)
Description: Safety population, defined as all participants who were randomized and received study treatment. All treatment-emergent serious adverse events are listed, whether or not they are related to study product.
Arm/Group | Fibrocaps + Gelatin Sponge | Gelatin Sponge
All-Cause Mortality (participants affected / at risk) | 8/480 | 2/239
Serious Adverse Events (participants affected / at risk) | 81/480 | 29/239
Other Adverse Events (participants affected / at risk) | 426/480 | 214/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrocaps + Gelatin Sponge (N=480) | Gelatin Sponge (N=239)
Pneumonia (Infections and infestations) | 4 | 2
Abdominal abscess (Infections and infestations) | 4 | 1
Postoperative wound infection (Infections and infestations) | 4 | 0
Sepsis (Infections and infestations) | 3 | 0
Wound infection (Infections and infestations) | 2 | 1
Abdominal sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Infectious peritonitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 3 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 2 | 2
Seroma (Injury, poisoning and procedural complications) | 2 | 2
Anastomotic leak (Injury, poisoning and procedural complications) | 2 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Small-for-size liver syndrome (Injury, poisoning and procedural complications) | 2 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 1 | 0
Pancreatic leak (Injury, poisoning and procedural complications) | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Ileus (Gastrointestinal disorders) | 3 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lymphorrhoea (Vascular disorders) | 3 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Silent myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac death (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Hernia obstructive (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Unintentional medical device removal by patient (General disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Hepatitis C antibody positive (Investigations) | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrocaps + Gelatin Sponge (N=480) | Gelatin Sponge (N=239)
Procedural Pain (Injury, poisoning and procedural complications) | 257 | 134
Nausea (Gastrointestinal disorders) | 120 | 48
Constipation (Gastrointestinal disorders) | 72 | 31
Incision site pain (Injury, poisoning and procedural complications) | 63 | 32
Hypotension (Vascular disorders) | 38 | 16
Anaemia (Blood and lymphatic system disorders) | 33 | 17
Insomnia (Psychiatric disorders) | 41 | 10
Pyrexia (General disorders) | 37 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 33 | 8
Hypertension (Vascular disorders) | 25 | 10
Vomiting (Gastrointestinal disorders) | 26 | 12
Procedural nausea (Injury, poisoning and procedural complications) | 22 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No